CLINICAL TRIAL: NCT04541511
Title: Comparison of the 6-minute Walking Test in a Corridor and on a Non-motorized Treadmill, Feasibility Study
Brief Title: Comparison of the 6-minute Walking Test in a Corridor and on a Non-motorized Treadmill
Acronym: TDM6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020_0047
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Walking, Difficulty
Keywords: 6-minutes walking test; 6-WT
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Intervention Model Description: * 31 healthy subjects
  * 6 patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subject (Experimental): Healthy subject will be asked to performed two 6-minutes walking test : one in a corridor and one on the non-motorized treadmill.
  Oxygen saturation, heart rate and Borg score will be collected before and after each test.
  Interventions: Diagnostic Test: 6-minutes walking test on a corridor; Diagnostic Test: 6-minutes walking test on a treadmill
- Patients (Experimental): Patients will be asked to to performed a 6-minutes walking test on the non-motorized treadmill and to answer a questionnaire regarding the acceptability and ease of use of the new method.
  Interventions: Diagnostic Test: 6-minutes walking test on a treadmill

INTERVENTIONS:
Diagnostic Test: 6-minutes walking test on a corridor — 6-minutes walking test on a corridor : patient will be asked to achieve the longest possible distance without running. He/she will be allowed to take breaks if he/she feels the need to do so.
  Arms: Healthy subject
Diagnostic Test: 6-minutes walking test on a treadmill — 6-minutes walking test on a treadmill : patient will be asked to achieve the longest possible distance without running on the treadmill. He/she will be allowed to take breaks if he/she feels the need to do so.

SUMMARY:
Evaluation of the equivalence of 6-minute walking test performed on a non-motorized treadmill to the reference test : a 6-minute walking test on a corridor.

DETAILED DESCRIPTION:
The Six-Minute Walk Test (6-WT) is a standardized test to assess a person's functional ability to walk as far as they can in six minutes. It is widely used in the assessment of functional disability in response to medical intervention in respiratory and cardiac conditions.

This test requires a corridor measuring between 20 and 30 metres and does not require any special technical equipment or training.

While the test appears simple to set up, factors such as the length or width of the corridor, and external disruptive elements, may affect the results. Indeed, the configuration of the test site plays a role in the test result. For example, the distance traveled in a 6-minute walking test is greater on a continuous circuit than in a lane that requires people to walk back and forth or when others are using the lane (zigzags, slowdowns). In a hospital setting, while it is easy to find a corridor that is long enough, it is not always possible to dedicate it exclusively to walking tests.

An alternative would be to perform this test on a non-motorized treadmill to avoid these biases. The main objective of this study is to evaluate the equivalence of a 6-minute walking test performed on a non-motorized treadmill to the reference test in healthy subjects. In addition, a small number of patients will be invited to perform a 6-minute CT scan on a non-motorized treadmill in order to first evaluate the perception and acceptability of this new method in this population (seniors, pathologies). If the results are conclusive, a similar study with patients only will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject 18 years of age or older
* Have signed a consent form
* Be affiliated with a Health Insurance Plan
* Having a pathology requiring the monitoring of the evolution of the distance performed by 6-WT (patients only)

Exclusion Criteria:

* Being unable to walk for several minutes for physical, neurological or psychological reasons
* Recent acute coronary syndrome
* Rest tachycardia greater than 120 pulses/min.
* Resting blood pressure greater than 180/100 mmHg
* Pregnant, Parturient or Nursing Women
* Persons deprived of liberty: minors or adults who are subject to a legal protection measure or who are unable to express their consent.
* Subjects under guardianship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2022-02-26 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
To assess the equivalence of walking distances obtained with the 6-minute walk test on a non-motorized treadmill to the baseline (6-WT on a corridor) test in healthy subjects. | [length on the test - 1 day]
  Total distance on the 6-WT on a corridor and on a non-motorized treadmill in healthy subjects.

SECONDARY OUTCOMES:
Evaluate the change in heart rate during the two test methods in healthy subjects | [length on the test - 1 day]
  Heart rate before and after each test : 6-WT on a corridor and on a non-motorized treadmill in healthy subjects.
Evaluate the change in oxygen saturation during the two test methods in healthy subjects. | [length on the test - 1 day]
  Oxygen saturation before and after each test : 6-WT on a corridor and on a non-motorized treadmill in healthy subjects.
To measure the perception of exertion after both test methods in healthy subjects. | [length on the test - 1 day]
  Borg scale before and after each test : 6-WT on a corridor and on a non-motorized treadmill in healthy subjects.
Evaluate patients' perception of the use of the new method. | [length on the test - 1 day]
  Non-standardized questionnaire assessing the acceptability and ease of use of the new method

CONTACTS AND LOCATIONS:
Overall Officials: Nina GOUDIER, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No